CLINICAL TRIAL: NCT01605136
Title: A Phase III, Multicentre, Double-Blind, Randomized, Placebo-Controlled Study to Confirm the Safety and Efficacy of Subcutaneous Bioresorbable Afamelanotide Implants in Patients With Erythropoietic Protoporphyria (EPP)
Brief Title: Phase III Confirmatory Study in Erythropoietic Protoporphyria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CUV039
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Erythropoietic Protoporphyria
Keywords: Erythropoietic Protoporphyria; EPP; Afamelanotide
MeSH Terms: conditions — Protoporphyria, Erythropoietic | interventions — afamelanotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Afamelanotide (Experimental): One 16mg subcutaneous implant every 2 months for 6 months.
  Interventions: Drug: Afamelanotide
- Placebo (Placebo Comparator): One placebo subcutaneous implant every 2 months for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Afamelanotide — One 16mg subcutaneous implant every 2 months for 6 months.
  Arms: Afamelanotide
Drug: Placebo — One placebo subcutaneous implant every 2 months for 6 months
  Arms: Placebo

SUMMARY:
This is a randomized placebo-controlled study to be conducted in two parallel study arms for a six month period (three doses). Between 75 and 100 eligible patients will be enrolled. Patients will receive afamelanotide (16 mg implants) or placebo according to the following dosing regimen:

* Group A will be administered afamelanotide implants on Days 0, 60 and 120
* Group B will be administered placebo implants on Days 0, 60 and 120

The number and severity of phototoxic reactions, the type and duration of sun exposure, treatment-emergent adverse events and the use of concomitant medication will be recorded by patients in study diaries between Days 0 and 180. Quality of life will be measured using the DLQI and EPP-QoL at Days 0, 60, 120 and 180. Participants will visit the clinic on Days 60, 120 and 180 for assessments of adverse events.

A subset of patients will be photoprovoked on the lower back and dorsal surface of the hand and the minimal symptom dose (MSD) will be determined on Days 0, 30, 60, 90 and 120.

DETAILED DESCRIPTION:
Afamelanotide is a man-made drug being studied for use as a preventative medication for Erythropoietic Protoporphyria (EPP) sufferers. It is a synthetically produced analogue of human alpha melanocyte stimulating hormone (alpha-MSH) and is available in Europe.

The purpose of this study is to look at the type and duration of sun exposure when patients are exposed to light. This study will also look at how the drug is tolerated when taken by people with EPP.

The study will involve the use of an implant, which comes in the form of a small rod to be administered under the skin. The implant may contain the study drug afamelanotide or a placebo (inactive medication).

Over 620 subjects have been treated with afamelanotide to date with no serious safety concerns identified. For this study, afamelanotide has been formulated as a controlled release depot injection (implant). This means that the afamelanotide will be released slowly into the body over a few days.

This study aims to confirm the photoprotective properties if afamelanotide demonstrated in the earlier Phase II and phase III studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with characteristic symptoms of EPP phototoxicity and a biochemically-confirmed diagnosis of EPP.
* Aged 18 years old and above (inclusive).
* Able to understand and sign the written Informed Consent Form.
* Willing to take precautions to prevent pregnancy until completion of the study (Day 180).

Exclusion Criteria:

* Any allergy to afamelanotide or the polymer contained in the implant or to lidocaine or other local anesthetic to be used during the administration of the study medication
* EPP patients with significant hepatic involvement
* Personal history of melanoma or dysplastic nevus syndrome.
* Current Bowen's disease, basal cell carcinoma, squamous cell carcinoma, or other malignant or premalignant skin lesions.
* Any other photodermatosis such as polymorphic light eruption, actinic prurigo, discoid lupus erythematosus, chronic actinic dermatitis or solar urticaria.
* Any evidence of clinically significant organ dysfunction or any clinically significant deviation from normal in the clinical or laboratory determinations.
* Acute history of drug or alcohol abuse (in the last 6 months).
* Patient assessed as not suitable for the study in the opinion of the Investigator (e.g. noncompliance history, allergic to local anesthetics, faints when given injections or giving blood).
* Participation in a clinical trial for an investigational agent within 30 days prior to the screening visit.
* Prior and concomitant therapy with medications which may interfere with the objectives of the study, including drugs that cause photosensitivity or skin pigmentation.
* Female who is pregnant (confirmed by positive serum β-HCG pregnancy test prior to baseline) or lactating.
* Females of child-bearing potential (pre-menopausal, not surgically sterile) not using adequate contraceptive measures (i.e. oral contraceptives, diaphragm plus spermicide, intrauterine device).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Desnick, MD, Principal Investigator — Mt. Sinai Medical Center
Locations (7):
- United States (7):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Henry Ford Medical Center, Detroit, Michigan
  - Mt. Sinai, New York, New York
  - Carolina's Medical Center Cannon Research, Charlotte, North Carolina
  - University of Texas, Galveston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Langendonk JG, Balwani M, Anderson KE, Bonkovsky HL, Anstey AV, Bissell DM, Bloomer J, Edwards C, Neumann NJ, Parker C, Phillips JD, Lim HW, Hamzavi I, Deybach JC, Kauppinen R, Rhodes LE, Frank J, Murphy GM, Karstens FPJ, Sijbrands EJG, de Rooij FWM, Lebwohl M, Naik H, Goding CR, Wilson JHP, Desnick RJ. Afamelanotide for Erythropoietic Protoporphyria. N Engl J Med. 2015 Jul 2;373(1):48-59. doi: 10.1056/NEJMoa1411481. PMID 26132941

RESULTS

PARTICIPANT FLOW:
Period: Study Period
Arm/Group | Afamelanotide | Placebo
Started | 48 | 45
Completed | 45 | 42
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 0 | 2
Period: Safety Follow-Up Period
Arm/Group | Afamelanotide | Placebo
Started | 45 | 42
Completed | 44 | 40
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Number of subjects enrolled into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afamelanotide | Placebo | Total
Number analyzed (Participants) | 48 | 45 | 93
Age, Continuous [Median (Full Range); unit: years] | 38.5 [20 to 65] | 35 [18 to 74] | 37 [18 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 44
  Male | 28 | 21 | 49

OUTCOME MEASURES:

1. Primary Outcome: Duration of Direct Sunlight Exposure Between 10:00 and 18:00 Hours on Days When no Pain Was Experienced (Pain Score of 0).
Description: The amount of direct sunlight exposure between 10:00 and 18:00 hours on days when no pain was experienced (e.g.11-point Likert pain score of 0). Time was recorded in a patient diary using 15 minute time blocks.
  The pain score is measured by the 11-point Likert Pain scale with minimum of 0 and maximum of 10.
  Likert Pain scale of 0 represents no pain and 10 represents worst imaginable pain.
Time Frame: Daily for 6 months
Population: Number of subjects (ITT population, from Patient Diary Card)
Measure: Median (Full Range); unit: hours
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 46 | 43
hours | 69.4 [0 to 650.50] | 40.8 [0.25 to 224.00]

2. Secondary Outcome: Combined Sun Exposure and Phototoxic Pain
Description: Time in direct sunlight exposure between 10:00 and 18:00 hours on days when no or mild pain was experienced (Likert scores of 0 to 3).
  The pain score is measured by the 11-point Likert Pain scale with minimum of 0 and maximum of 10.
  Likert Pain scale of 0 represents no pain and 10 represents worst imaginable pain.
Time Frame: Daily for 6 months
Population: Number of subjects (ITT population, from Patient Diary Card)
Measure: Median (Full Range); unit: hours
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 46 | 43
hours | 80.0 [0.5 to 825.0] | 51.0 [1.25 to 251.0]

3. Secondary Outcome: Sun Exposure
Description: Duration of direct sunlight exposure between 10:00 and 18:00 hours during the study.
Time Frame: Daily for 6 months
Population: Number of subjects (ITT population, from Patient Diary Card)
Measure: Median (Full Range); unit: hours
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 46 | 43
hours | 83.50 [0.50 to 825.00] | 65.25 [3.50 to 278.50]

4. Secondary Outcome: Quality of Life Score
Description: The Quality of life of participant is measured using DLQI and EPP QoL. The Dermatology Life Quality Index (DLQI) is a simple practical measure for routine clinical use.
  The DLQI ranges from 0 (no impact on life) to 30 (significant impact on life) . The Erthropoietic protoporphyria quality of life measure (EPP-QoL) scores range from 0 (worst imaginable QoL) to 100 (best possible QoL).
Time Frame: Day 60, Day 120, and Day 180 or early termination.
Population: The number of participants analyzed differs from the overall number of participants analyzed because the data was either incomplete and/or missing. Only data from those who completed the Quality of Life assessments are included at each time point.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 47 | 43
units on a scale
  DLQI - Day 0 (baseline): number analyzed (Participants) | 46 | 43
  DLQI - Day 0 (baseline) | 10.0 [0 to 26] | 11.0 [0 to 22]
  DLQI - Day 60: number analyzed (Participants) | 46 | 43
  DLQI - Day 60 | 2.0 [0 to 21] | 4.0 [0 to 21]
  DLQI - Day 120: number analyzed (Participants) | 45 | 42
  DLQI - Day 120 | 0.5 [0 to 16] | 2.5 [0 to 19]
  DLQI - Day 180/Early Termination: number analyzed (Participants) | 46 | 43
  DLQI - Day 180/Early Termination | 1.0 [0 to 16] | 1.0 [0 to 14]
  EPP QOL - Day 0 (baseline) | 19.4 [0 to 83] | 22.2 [3 to 81]
  EPP QOL - Day 60 | 77.8 [0 to 100] | 55.6 [6 to 97]
  EPP QOL - Day 120: number analyzed (Participants) | 46 | 42
  EPP QOL - Day 120 | 81.9 [17 to 100] | 61.1 [6 to 97]
  EPP QOL - Day 180/Early Termination: number analyzed (Participants) | 46 | 43
  EPP QOL - Day 180/Early Termination | 86.1 [6 to 100] | 69.4 [11 to 100]

5. Secondary Outcome: Photoprovocation
Description: A subset of subjects was photoprovoked on the dorsal surface of the hand (predilection place) and lower back and the minimum symptom dose (MSD) determined on Days 0, 30, 60, 90 and 120.
  The amount of radiation required to provoke the first clinical symptom was recorded.
Time Frame: Day 0, Day 30, Day 60, Day 90 and Day 120.
Measure: Median (Full Range); unit: J/cm^2
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 10 | 10
J/cm^2
  Day 0: dorsal surface of the hand | 48.9 [2.3 to 172] | 21.0 [1.1 to 200]
  Change at Day 30: dorsal surface of the hand | 197.5 [6.4 to 291] | 75.6 [-42.7 to 292]
  Change at Day 60: dorsal surface of the hand | 128.3 [-62.8 to 298] | 36.3 [-1.5 to 157]
  Change at Day 90: dorsal surface of the hand | 208.3 [41.6 to 298] | 13.9 [-51.3 to 289]
  Change at Day 120: dorsal surface of the hand | 162.1 [22.9 to 291] | 1.9 [-54.3 to 289]
  Day 0: lower back | 32.0 [2.1 to 157] | 24.1 [3.7 to 300]
  Change at Day 30: lower back | 237.1 [9.1 to 285] | 44.8 [-103.8 to 294]
  Change at Day 60: lower back | 50.7 [-56.4 to 285] | 4.3 [-210.3 to 124]
  Change at Day 90: lower back | 227.5 [96.0 to 298] | -2.4 [-132.6 to 124]
  Change at Day 120: lower back | 82.5 [10.0 to 271] | 12.1 [-187.4 to 124]

6. Secondary Outcome: Maximum Severity of Phototoxic Reaction Experienced by Participants
Description: The phototoxicity - phototoxic pain secondary endpoint has been divided into two secondary outcome measures.
  The days on which the participant experienced pain as a result of phototoxic reactions (caused by exposure to natural light) was recorded in a study diary. On each day such a reaction occurred, the participant scored the level of pain using an 11-point Likert pain scale, with minimum of 0 and maximum of 10. The 11-point Likert pain scale with a value of 0 represents no pain and 10 represents worst imaginable pain.
  The maximum severity of a phototoxic reaction was determined by the highest daily 11-point Likert scale score that occurred during that phototoxic reaction.
Time Frame: Daily for 6 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 46 | 43
score on a scale | 4.0 [0 to 8] | 5.0 [0 to 9]

7. Secondary Outcome: Total Number Phototoxic Reactions Experienced by Participants
Description: The phototoxicity - phototoxic pain secondary endpoint has been divided into two secondary outcome measures.
  The number of episodes was the endpoint. The days on which the participant experienced pain as a result of phototoxic reactions (caused by exposure to natural light) was recorded in a study diary. On each day such a reaction occurred, the participant scored the level of pain using an 11-point Likert pain scale, with minimum of 0 and maximum of 10. The 11-point Likert Pain scale with a value of 0 represents no pain and 10 represents worst imaginable pain.
  The number of phototoxic reactions was determined by counting the number of episodes on which participants report a 11-point Likert scale score of 4 or more for one or more consecutive days.
Time Frame: Daily for 6 months
Measure: Median (Full Range); unit: episodes
Arm/Group | Afamelanotide | Placebo
Number analyzed (Participants) | 46 | 43
episodes | 4 [0 to 196] | 6 [0 to 507]

ADVERSE EVENTS:
Time Frame: Visit 1 (Day 0) - Visit 4 (Day 180)
Arm/Group | Afamelanotide | Placebo
Serious Adverse Events (participants affected / at risk) | 3/48 | 2/45
Other Adverse Events (participants affected / at risk) | 45/48 | 39/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afamelanotide (N=48) | Placebo (N=45)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Melanocytic naevus (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afamelanotide (N=48) | Placebo (N=45)
Nausea (Gastrointestinal disorders) | 9 | 8
Pain (General disorders) | 4 | 4
Nasopharyngitis (Infections and infestations) | 6 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Headache (Nervous system disorders) | 19 | 13
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Implant site discolouration (General disorders) | 9 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Fatigue (General disorders) | 3 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 3
Influenza (Infections and infestations) | 2 | 7
Sinusitis (Infections and infestations) | 3 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Migraine (Nervous system disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No